CLINICAL TRIAL: NCT03016637
Title: Pancreatic Core Biopsy Needle Study (PANCOBE)
Brief Title: Pancreatic Core Biopsy Needle Study in Patients Suspected of Pancreatic Malignancy
Acronym: PANCOBE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Michael Bau Mortensen, Professor, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MBM-71
Record Dates: First submitted 2017-01-09; First posted 2017-01-10 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Pancreatic Cancer
Keywords: endoscopic ultrasonography; EUS-FNA
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EUS biopsy (Experimental): EUS guided SharkCore (TM) biopsy of pancreatic lesions suspected of malignancy
  Interventions: Device: SharkCore (TM) FNB Exchange System

INTERVENTIONS:
Device: SharkCore (TM) FNB Exchange System
  Other Names: 25 Gauge or 22 Gauge SharkCore needle

SUMMARY:
This study evaluates whether a new endoscopic ultrasonography (EUS) histology needle may improve the diagnostic yield during biopsies of pancreatic lesions

DETAILED DESCRIPTION:
Pancreatic cancer has a poor prognosis, and a quick and correct diagnosis is essential. Endoscopic ultrasonography (EUS) is highly accurate regarding the detection of pancreatic cancer, and EUS guided fine-needle aspiration biopsy (EUS-FNA) may be used to verify the diagnosis in patients with non-resectable or metastatic disease. However, EUS-FNA is only diagnostic in approximately 70% of the cases, and the reported number of "atypical", "suspicious" and "insufficient" biopsies varies.

SharkCore (TM) is a new type of EUS fine needle that allows the extraction of macroscopic tissue fractions ("trucut biopsies") instead of single cells or cluster of cells. Preliminary data suggest that EUS guided trucut biopsies from the pancreatic lesions are technically feasible without increasing the number of complications.

This prospective study evaluates the clinical outcome and potential complications following EUS guided biopsy of pancreatic lesions suspected of cancer using a 25 Gauge or 22 Gauge SharkCore needle.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic lesion suspected of malignancy and EUS biopsy indicated

Exclusion Criteria:

* Resectable pancreatic lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of conclusive biopsies | minimum 6 moths after biopsy

SECONDARY OUTCOMES:
Complications | 2 weeks after biopsy
  All contacts to the secondary health care system
Quality test of biopsies | 2 weeks after biopsy
  Biopsies divided into:
  1) diagnostic 2a) if not diagnostic - representative material 2b) if not diagnostic - not representative material 3) Insufficient material

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Mortensen, Professor, Study Director — Odense University Hospital, University of Southern denmark
Locations (1):
- Odense University Hospital, Odense, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hewitt MJ, McPhail MJ, Possamai L, Dhar A, Vlavianos P, Monahan KJ. EUS-guided FNA for diagnosis of solid pancreatic neoplasms: a meta-analysis. Gastrointest Endosc. 2012 Feb;75(2):319-31. doi: 10.1016/j.gie.2011.08.049. PMID 22248600
- [Background] Bardales RH, Stelow EB, Mallery S, Lai R, Stanley MW. Review of endoscopic ultrasound-guided fine-needle aspiration cytology. Diagn Cytopathol. 2006 Feb;34(2):140-75. doi: 10.1002/dc.20300. PMID 16511852
- [Background] Iglesias-Garcia J, Poley JW, Larghi A, Giovannini M, Petrone MC, Abdulkader I, Monges G, Costamagna G, Arcidiacono P, Biermann K, Rindi G, Bories E, Dogloni C, Bruno M, Dominguez-Munoz JE. Feasibility and yield of a new EUS histology needle: results from a multicenter, pooled, cohort study. Gastrointest Endosc. 2011 Jun;73(6):1189-96. doi: 10.1016/j.gie.2011.01.053. Epub 2011 Mar 21. PMID 21420083
- [Background] Bang JY, Hebert-Magee S, Trevino J, Ramesh J, Varadarajulu S. Randomized trial comparing the 22-gauge aspiration and 22-gauge biopsy needles for EUS-guided sampling of solid pancreatic mass lesions. Gastrointest Endosc. 2012 Aug;76(2):321-7. doi: 10.1016/j.gie.2012.03.1392. Epub 2012 May 31. PMID 22658389
- [Background] Mortensen MB, Fristrup C, Holm FS, Pless T, Durup J, Ainsworth AP, Nielsen HO, Hovendal C. Prospective evaluation of patient tolerability, satisfaction with patient information, and complications in endoscopic ultrasonography. Endoscopy. 2005 Feb;37(2):146-53. doi: 10.1055/s-2005-861142. PMID 15692930